CLINICAL TRIAL: NCT03408886
Title: Microbiota Transfer Therapy for Adults With Autism Spectrum Disorder (ASD) Who Have Gastrointestinal Disorders
Acronym: MTT-ASD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTT-Adults-1; Wi1XWH-16-1-0492 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Autism Spectrum Disorder; Gastrointestinal Disorder
Keywords: fecal transplant; fecal microbiota transplant; microbiota transplant; vancomycin; moviprep
MeSH Terms: conditions — Autism Spectrum Disorder; Gastrointestinal Diseases | interventions — Vancomycin; MoviPrep; Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: There are two groups. In Part 1, group A receives treatment and group B receives placebo. In Part 2, group A continues to receive treatment, and group B is switched to treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In Part 1, everyone is blinded except for the research pharmacist. In Part 2, the participants and study coordinator are unblinded, but the professional evaluators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A receives treatment in Part 1 and Part 2
  Interventions: Drug: Vancomycin; Drug: MoviPrep; Biological: Full Spectrum Microbiota
- Group B (Other): Group B receives no treatment in Part 1, but does receive treatment in Part 2
  Interventions: Drug: MoviPrep; Biological: Full Spectrum Microbiota

INTERVENTIONS:
Drug: Vancomycin — Oral vancomycin is administered to reduce pathogenic bacteria.
  Arms: Group A
Drug: MoviPrep — MoviPrep is given at the end of vancomycin therapy to remove the vancomycin and remaining bacteria prior to administering Full-Spectrum Microbiota
Biological: Full Spectrum Microbiota — Gut bacteria from healthy human donors are administered orally in a pill form
  Other Names: fecal microbiota transplant

SUMMARY:
This is a clinical trial of Microbiota Transplant Therapy (MTT) for adults with autism spectrum disorders (ASD) who have gastrointestinal problems.

Previous research has shown that individuals with ASD have a low diversity of gut bacteria, and low diversity is generally associated with poor gastrointestinal (GI) health. We previously found that MTT therapy for children with ASD and GI symptoms was helpful in reducing their GI symptoms, reducing their ASD symptoms, and increasing their diversity of gut bacteria.

This clinical trial will investigate the hypothesis that MTT therapy will be helpful for adults with ASD who have GI symptoms.

DETAILED DESCRIPTION:
For adults ages 18-60 years with ASD and gastrointestinal problems, the investigators propose a Phase 2 clinical trial to evaluate the safety and efficacy of MTT. The study will also determine if longer treatment is beneficial, and to conduct a longer observation after treatment stops to determine long-term safety and efficacy. The three parts of this trial are described below.

Part 1: Placebo-Controlled Treatment The trial will begin with a randomized, double-blind, placebo-controlled trial which will include a 2-week treatment with oral vancomycin (or placebo), then 1 day of Moviprep to cleanse the bowel of vancomycin and bacteria/feces (all participants, since its bowel-emptying effect cannot be blinded), followed by oral administration of Full Spectrum Microbiota (FSM) or placebo. An initial high dose of FSM (or placebo) for two days will be followed by a lower maintenance dose of FSM (or placebo) for 8 weeks.

Part 2 Extension and Cross-Over

* For the treatment group from Part 1, there will be an 8-week extension of the maintenance dose, to determine if longer treatment has additional benefits.
* For the placebo group from Part 1, they will receive MoviPrep, an initial high dose of FSM for 2 days, and then a lower dose of FSM for 8 weeks (similar to the treatment group in Part 1, but without the vancomycin). This will help us determine if pre-treatment with vancomycin is needed or not.

Part 3: Follow-up There will be follow-up evaluations at 6, 12, and 18 months after treatment is stopped, to assess long-term efficacy and possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18-60 years
2. Diagnosis of autism per both the Autism Diagnostic Interview - Revised (ADI-R) and the Childhood Autism Rating Scale 2 (CARS-2).
3. GI disorder as defined below that has lasted for at least 3 years.
4. No changes in medications, supplements, diet, therapies, or education in last 3 months, and no intention to change them during the clinical trial.
5. General good physical health aside from gastrointestinal problems
6. Neurotypical adult observer (such as parent, guardian, or sibling) who observes adult for at least 4 hours/week who can serve as an Evaluator to complete questionnaires on their symptoms with the assistance of the Participant as much as they are able.
7. Ability to swallow pills (without chewing)

Exclusion Criteria:

1. Antibiotics in last 3 months
2. Probiotics in last 2 months, or fecal transplant in last 12 months
3. Single-gene disorder (Fragile X, etc.)
4. Major brain malformation
5. Tube feeding
6. Severe gastrointestinal problems that require immediate treatment (life-threatening)
7. Ulcerative Colitis, Crohn's Disease, diagnosed Celiac Disease, Eosinophilic Gastroenteritis, or similar conditions
8. Severely underweight/malnourished
9. Recent or scheduled surgeries
10. Current participation in other clinical trials
11. Females who are pregnant or who are sexually active without effective birth control. We will conduct a urine pregnancy test on all female participants as part of the screening and at each clinical visit.
12. Allergy or intolerance to vancomycin or MoviPrep
13. Clinically significant abnormalities at baseline on two blood safety tests: Comprehensive Metabolic Panel and Complete Blood Count with Differential.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Childhood Autism Rating Scale (CARS) from baseline to 10 weeks | baseline; month 2.5, 4.5, 10.5, 16.5, 22.5
  An evaluation by a trained evaluator of autism symptoms. The range is 15-60, and scores in the range of 27-30 or higher are indicative of autism.

SECONDARY OUTCOMES:
Change in Daily Stool Log (DSL) from baseline to 10 weeks | baseline for 2 weeks; daily for 18 weeks, and 2 weeks at month 10, 16, 22
  The DSL is a report of the number and type of stools over 14 days. Each stool is rated on a scale of 1-7, where 1=very hard, 4=normal, 7=very soft/liquid. The DSL is scored by the number of days of an abnormal stool (type 1-2 or 6-7) or no stool.
Change in Social Responsiveness Scale - 2 from baseline to 10 weeks of treatment | baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18; months 10.5, 16.5, 22.5
  A questionnaire about social skills, where higher scores suggest more severe autism. Scores range from 0 to 195, with higher scores indicating more severe problems.
Change in Aberrant Behavior Checklist from baseline to 10 weeks | baseline; month 2.5, 4.5, 10.5, 16.5, 22.5
  a questionnaire about aberrant behaviors. Scores range from 0 to 174, with higher scores indicating more severe behaviors

OTHER OUTCOMES:
Change in Gastrointestinal Stool and Symptom Questionnaire for Autism, from baseline to 10 weeks | baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18; month 10.5, 16.5, 22.5
  a questionnaire about GI-related symptoms.
Change in Microbiome composition from baseline to 10 weeks | baseline; month 1, 2.5, 3.5, 4.5, 10.5, 16.5, 22.5
  analysis of the bacterial composition of stool samples, at the species, genus, and phylum level
Change in the Vineland Adaptive Behavior Scale - II, from baseline to 10 weeks | baseline; month 2.5, 4.5, 22.5
  questionnaire about adaptive behaviors; it yields the developmental age of the participant
Change in Ohio State University Clinical Impressions Scale, from baseline 10 weeks | baseline; month 2.5, 4.5
  assessment of autism symptoms by a clinician. It rates 10 symptoms on a scale of 1-7, with higher scores indicating worse symptoms.
Change in Parent Global Impressions, from baseline to 10 weeks | baseline; weeks 2, 4, 6, 8, 10, 12, 14, 16, 18; month 10.5, 16.5, 22.5
  Assessment of autism symptoms. It rates 20 symptoms on a scale of 1-7, with higher scores indicating worse symptoms

CONTACTS AND LOCATIONS:
Overall Officials: James B Adams, PhD, Study Director — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang DW, Adams JB, Gregory AC, Borody T, Chittick L, Fasano A, Khoruts A, Geis E, Maldonado J, McDonough-Means S, Pollard EL, Roux S, Sadowsky MJ, Lipson KS, Sullivan MB, Caporaso JG, Krajmalnik-Brown R. Microbiota Transfer Therapy alters gut ecosystem and improves gastrointestinal and autism symptoms: an open-label study. Microbiome. 2017 Jan 23;5(1):10. doi: 10.1186/s40168-016-0225-7. PMID 28122648
- See also: link to more information about the research group — http://autism.asu.edu